CLINICAL TRIAL: NCT02755129
Title: FRailty WAlking Patterns (FRAP) Study
Acronym: FRAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic BRC (Industry)
Collaborators: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FRAP1
Record Dates: First submitted 2016-03-02; First posted 2016-04-28 (Estimated); Results first posted 2020-03-25 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- single arm (Other): Single arm, all the patients enrolled will perform the same walking exercises.
  On arrival to the rehabilitation center subjects will have the Reveal LINQ, the 3D-accelerometers (one on the chest by medical-grade adhesives and a second at the level of the waist over the top of a medical grade adhesive) and the Holter attached externally. Then, they will be asked to perform the following exercises:
  * Walking Exercises-4 Meter Gait Speed (4MGS) Test Walking exercises - Six Minute Walk (6MW) Test
  * Walking exercises - 4 Meter Gait Speed (4MGS) Test
  * Walking Exercises - Five Times Sit to Stand (FTSTS) Test
  * Walking Exercises - Expanded Timed Get-Up-and-Go (ETGUG) Test
  Interventions: Other: Walking Exercises-Six Minute Walk (6MW) Test; Other: Walking Exercises-4 Meter Gait Speed (4MGS) Test; Other: Walking Exercises-Five Times Sit to Stand (FTSTS) Test; Other: Walking Exercises-Expanded Timed Get-Up-and-Go (ETGUG) Test; Other: Reveal LINQ accelerometer; Other: 3D accelerometer

INTERVENTIONS:
Other: Walking Exercises-Six Minute Walk (6MW) Test — The Six Minute Walk (6MW) Test measures the distance an individual is able to walk over a total of six minutes on a flat surface. The goal is for the individual to walk as far as possible in six minutes. The Six Minute Walk (6MW) test will be performed within the Computer Assisted Rehabilitation Environment (CAREN) system system environment - single arm
Other: Walking Exercises-4 Meter Gait Speed (4MGS) Test — The 4 Meter Gait Speed (4MGS) Test measures the gait speed an individual is able to walk over 4 meters on a flat surface. The goal is for the individual to walk as fast as possible over 4 meters.
  It will be repeated 3 times within the aforementioned 6MW test (after approximately 1, 3 and 5 minutes) to get variability due to subject tiredness. The test will be performed within the CAREN system environment. - single arm
Other: Walking Exercises-Five Times Sit to Stand (FTSTS) Test — The Five Times Sit to Stand (FTSTS) Test measures the time a subject takes to stand up from an armchair 5 times in a row, without stopping in between. It is a short test which measures dynamic balance and functional mobility - single arm
Other: Walking Exercises-Expanded Timed Get-Up-and-Go (ETGUG) Test — The Expanded Timed Get-Up-and-Go (ETGUG) Test measures the time it takes a subject to stand up from an armchair, walk a distance of 10 m, turn, walk back to the chair, and sit down. It is a short test of basic mobility skills for frail community-dwelling elderly. - single arm
Other: Reveal LINQ accelerometer — Walking exercises test
Other: 3D accelerometer — Walking exercises test

SUMMARY:
The aim of this study is to evaluate sit-stand phases and gait speed detection using an externally worn Reveal LINQ (TM) compared to an external reference (3D accelerometer, and/or the Computer Assisted Rehabilitation Environment (CAREN) system) in one center in the Netherlands

DETAILED DESCRIPTION:
Frailty is a geriatric syndrome characterized by reduced homeostatic reserves, exposing the organism to extreme vulnerability to endogenous and exogenous stressors.

Frailty is prevalent in older people and involves a progressive physiological decline of multiple body systems, typical signs and symptoms include weight loss, fatigue, muscle weakness, slow or unsteady gait declines in activity.

Frailty is increasingly recognized as an important prognostic indicator in heart failure (HF) and is more prevalent in HF than the general population.

The identification of frailty in its early stage is important because interventions may potentially prevent, or delay the clinical consequences of frailty.

Of particular focus in this study will be walking speed as prior research has demonstrated that slow gait speed has the strongest prognostic ability of the traditional components used to assess frailty, and has been reported as one of the strongest to predict adverse outcomes, such as mobility disability, falls, or hospitalization.

Also of interest is the detection of posture changes as this may have implications for detecting changes in sleeping habits and could also provide context for other biomarker signals collected by the LINQ device.

The literature has been reviewed and the scientific soundness of the proposed analytical techniques evaluated. The rationale for this study design is to evaluate the feasibility of using the Reveal LINQ™ to monitoring walking patterns.

HF patients (the target population for the study in discussion) would make it possible to test the sensitivity of the accelerometer embedded in the LINQ device in a small cohort of subjects with reduced mobility and for which frailty is more prevalent than the general population, as well as recognized as an important prognostic indicator.

No risk to the subjects is expected with this study.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Heart Failure in New York Heart Association (NHYA) class II and class III
* Willing to sign the informed consent form.
* At least 18 years of age.

Exclusion Criteria:

* • Not able to walk continuously for a period of 6 minutes and perform the walking exercises as necessary for the study protocol.

  * Any known allergy to Titanium
  * Any concomitant conditions which in the opinion of the investigator would not allow accurate measurement of gait and frailty parameters with an externally worn device.
  * Any concomitant condition which in the opinion of the investigator would not allow a safe participation in the study.
  * Enrolled in another study that could confound the results of this study, without documented pre-approval from a Medtronic study manager.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-09-20 (Actual); Primary Completion 2017-04-20 (Actual); Study Completion 2017-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Meijer,, Principal Investigator — Maastricht University
Locations (1):
- NUTRIM School of Nutrition and Translational Research in Metabolism of the Faculty Health, Medicine and Life Sciences, Maastricht University,, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- All Study Participants: Patients with Chronic Heart Failure. No control group has been used for this study, but all the patients enrolled will perform the same walking exercises.
  On arrival to the rehabilitation center subjects will have the Reveal LINQ, the 3D-accelerometers (one on the chest by medical-grade adhesives and a second at the level of the waist over the top of a medical grade adhesive) and the Holter attached externally. Then, they will be asked to perform the following exercises:
  * Walking exercises - Six Minute Walk (6MW) Test
  * Walking exercises - 4 Meter Gait Speed (4MGS) Test
  * Walking Exercises - Five Times Sit to Stand (FTSTS) Test
  * Walking Exercises - Expanded Timed Get-Up-and-Go (ETGUG) Test
Period: Overall Study
Arm/Group | All Study Participants
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Patients with Chronic Heart Failure. No control group has been used for this study, but all the patients enrolled will perform the same walking exercises.
  On arrival to the rehabilitation center, subjects will have the Reveal LINQ, the 3D-accelerometers (one on the chest by medical-grade adhesives and a second at the level of the waist over the top of a medical grade adhesive) and the Holter attached externally. Then, they will be asked to perform the following exercises:
  * Walking exercises - Six Minute Walk (6MW) Test
  * Walking exercises - 4 Meter Gait Speed (4MGS) Test
  * Walking Exercises - Five Times Sit to Stand (FTSTS) Test
  * Walking Exercises - Expanded Timed Get-Up-and-Go (ETGUG) Test
Arm/Group | All Study Participants
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Netherlands | 15

OUTCOME MEASURES:

1. Primary Outcome: Correlation of Gait Speed Between Reveal LINQ Accelerometer, Validation Accelerometer and/or Computer Assisted Rehabilitation System by Walking Exercises
Description: The gait speed will be calculated from the Reveal LINQ accelerometer signals, from the validation accelerometer and / or from the computer assisted rehabilitation system during the walking exercises.
  We will calculate the average correlation coefficient over all patients and exercises.
  It is reported as score on a scale, with minimum value= -1 and maximum value = 1.
  Higher absolute values mean higher correlation.
Time Frame: During walking exercises visit, 1 Day
Population: 15 subjects were enrolled and completed the study. All subjects met the inclusion and exclusion criteria.
  One subject did not have readable device data and as such was excluded from the analysis.
Measure: Number; unit: Correlation Coefficient
Groups:
- Correlation Coefficient - Six Minute Walk (6MW) Test: Patients with Chronic Heart Failure. No control group used. All patients enrolled performed the same walking exercises. On arrival to the rehabilitation center subjects will have the Reveal LINQ, the 3D-accelerometers (one on the chest by medical-grade adhesives and a second at the level of the waist over the top of a medical grade adhesive) and the Holter attached externally. Then, the correlation coefficient for gait speed across devices for Six Minute Walk (6MW) Test is calculated.
- Correlation Coefficient - 4 Meter Gait Speed (4MGS) Test: Patients with Chronic Heart Failure. No control group used. All patients enrolled performed the same walking exercises. On arrival to the rehabilitation center subjects will have the Reveal LINQ, the 3D-accelerometers (one on the chest by medical-grade adhesives and a second at the level of the waist over the top of a medical grade adhesive) and the Holter attached externally. Then, the correlation coefficient for gait speed across devices for 4 Meter Gait Speed (4MGS) Test is calculated.
- Correlation Coefficient - Five Times Sit to Stand (FTSTS) Test: Patients with Chronic Heart Failure. No control group used. All patients enrolled performed the same walking exercises. On arrival to the rehabilitation center subjects will have the Reveal LINQ, the 3D-accelerometers (one on the chest by medical-grade adhesives and a second at the level of the waist over the top of a medical grade adhesive) and the Holter attached externally. Then, the correlation coefficient for gait speed across devices for Five Times Sit to Stand (FTSTS) Test is calculated.
- Correlation Coefficient - ETGUG Test: Patients with Chronic Heart Failure. No control group used. All patients enrolled performed the same walking exercises. On arrival to the rehabilitation center subjects will have the Reveal LINQ, the 3D-accelerometers (one on the chest by medical-grade adhesives and a second at the level of the waist over the top of a medical grade adhesive) and the Holter attached externally. Then, the correlation coefficient for gait speed across devices for Expanded Timed Get-Up-and-Go (ETGUG) Test is calculated.
Arm/Group | Correlation Coefficient - Six Minute Walk (6MW) Test | Correlation Coefficient - 4 Meter Gait Speed (4MGS) Test | Correlation Coefficient - Five Times Sit to Stand (FTSTS) Test | Correlation Coefficient - ETGUG Test
Number analyzed (Participants) | 14 | 14 | 14 | 14
Correlation Coefficient
  Correlation per each Exercise | 0.97 | 0.93 | 0.86 | 0.91
  Average Correlation Across All Exercises | 0.91 | 0.91 | 0.91 | 0.91
Statistical Analysis 1: Comparison: Correlation Coefficient - Six Minute Walk (6MW) Test vs Correlation Coefficient - 4 Meter Gait Speed (4MGS) Test vs Correlation Coefficient - Five Times Sit to Stand (FTSTS) Test vs Correlation Coefficient - ETGUG Test; Test type: Other; To assess the similarity between the Reveal LINQ measures and those from the reference system, correlation coefficients were used. The correlation coefficient was calculated over windows of 4 seconds and averaged for each exercise. Then, the average correlation coefficient over all patients and exercise was calculated

ADVERSE EVENTS:
Time Frame: No adverse event collected in this study
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed
Arm/Group | All Study Participants
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-02-17): https://cdn.clinicaltrials.gov/large-docs/29/NCT02755129/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-20): https://cdn.clinicaltrials.gov/large-docs/29/NCT02755129/SAP_001.pdf